CLINICAL TRIAL: NCT06620432
Title: High Segmental Hysterotomy Vs. Low Segmental Hysterotomy: Association with the Incidence of Uterine Wall Defects After Cesarean Section
Brief Title: High Vs. Low Segmental Hysterotomy: Impact on Uterine Wall Defects Post-Cesarean
Acronym: HISEAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024.079
Record Dates: First submitted 2024-08-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Placenta Accreta Spectrum
Keywords: High segmental hysterotomy; Low segmental hysterotomy; Caesarean section; hysterotomy defects
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low Segment Hysterotomy + Crossed hysterorrhaphy (Active Comparator): The participant will undergo a cesarean section in which the surgical technique of Low Segment Hysterotomy and Crossed hysterorrhaphy for uterine closure will be employed. The initial incision and skin closure will be performed at the discretion of the gynecologist.
  Interventions: Procedure: Low segment hysterotomy; Procedure: Crossed hysterorrhaphy
- High Segment Hysterotomy + Crossed hysterorrhaphy (Experimental): The participant will undergo a cesarean section in which the surgical technique of High Segment Hysterotomy and Crossed hysterorrhaphy for uterine closure will be employed. The initial incision and skin closure will be performed at the discretion of the gynecologist.
  Interventions: Procedure: High segment hysterotomy; Procedure: Crossed hysterorrhaphy
- Low Segment Hysterotomy + Non-Crossed hysterorrhaphy (Experimental): The participant will undergo a cesarean section in which the surgical technique of Low Segment Hysterotomy and Non-Crossed hysterorrhaphy for uterine closure will be employed. The initial incision and skin closure will be performed at the discretion of the gynecologist.
  Interventions: Procedure: Low segment hysterotomy; Procedure: Non-Crossed hysterorrhaphy
- High Segment Hysterotomy + Non-Crossed hysterorrhaphy (Experimental): The participant will undergo a cesarean section in which the surgical technique of High Segment Hysterotomy and Non-Crossed hysterorrhaphy for uterine closure will be employed. The initial incision and skin closure will be performed at the discretion of the gynecologist.
  Interventions: Procedure: High segment hysterotomy; Procedure: Non-Crossed hysterorrhaphy

INTERVENTIONS:
Procedure: Low segment hysterotomy — A low segment hysterotomy is a surgical procedure in which an incision is made in the lower segment of the uterus, typically during a cesarean section or other uterine surgeries. This approach is preferred because the lower uterine segment is thinner and less vascular, reducing the risk of bleeding and complications during and after the procedure. The incision is typically horizontal.
  Arms: Low Segment Hysterotomy + Crossed hysterorrhaphy; Low Segment Hysterotomy + Non-Crossed hysterorrhaphy
Procedure: High segment hysterotomy — A high segment hysterotomy is a surgical procedure involving an incision in the upper segment of the uterus.
  Arms: High Segment Hysterotomy + Crossed hysterorrhaphy; High Segment Hysterotomy + Non-Crossed hysterorrhaphy
Procedure: Crossed hysterorrhaphy — Crossed hysterorrhaphy is a surgical technique used to close the uterine incision following a hysterotomy, particularly during cesarean sections. In this method, the sutures are placed in a crossed or X-shaped pattern, which helps to evenly distribute tension across the incision site.
  Arms: High Segment Hysterotomy + Crossed hysterorrhaphy; Low Segment Hysterotomy + Crossed hysterorrhaphy
Procedure: Non-Crossed hysterorrhaphy — Non-crossed hysterorrhaphy is a surgical technique used to close a uterine incision, typically after a hysterotomy, such as during a cesarean section. In this method, the sutures are placed in a linear, parallel fashion rather than in a crossed or X-shaped pattern
  Arms: High Segment Hysterotomy + Non-Crossed hysterorrhaphy; Low Segment Hysterotomy + Non-Crossed hysterorrhaphy

SUMMARY:
The purpose of this clinical trial is to compare the incidence of defects in the uterine wall at the site of the scar (niche) and surgical complications when using high-segment versus low-segment hysterotomy, with both cross-suturing and non-cross-suturing techniques, in pregnant patients undergoing their first cesarean section.

Researchers will compare four arms:

* Low Segment Hysterotomy + Crossed hysterorrhaphy
* High Segment Hysterotomy + Crossed hysterorrhaphy
* Low Segment Hysterotomy + Non-Crossed hysterorrhaphy
* High Segment Hysterotomy + Non-Crossed hysterorrhaphy

Participants will:

* Cesarean delivery
* Attend a follow up appointment between 6 to 16 weeks post surgery where will be perform a transvaginal sonography.

DETAILED DESCRIPTION:
This study will be conducted as a single-blind trial. Patients will be approached in the delivery room, where a comprehensive review of the inclusion and exclusion criteria checklist will be conducted to determine their eligibility for the study. Once eligible patients are identified, the study will be thoroughly explained to them, highlighting its purpose, potential benefits, and risks. This will be followed by a detailed discussion of the informed consent form to ensure that participants fully understand what their involvement entails.

Upon obtaining informed consent, a randomization process will be implemented to allocate participants to one of the four study arms. The assigned procedure will be performed by their attending gynecologist, who is familiar with their medical history and care needs. Throughout the study, various outcomes will be measured, including intraoperative findings, postoperative recovery, and post-discharge progress.

A transvaginal pelvic ultrasound will be ordered to be performed between 6 and 16 weeks postoperatively. During the single follow-up appointment, this imaging evaluation will be carried out to determine the presence or absence of an isthmocele, as well as to assess its characteristics, such as size and location, if present.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged ≥ 18 years.
* Confirmed pregnancy through clinical history or ultrasound between 36 and 42 weeks of gestation.
* Indication by the attending gynecologist for a first cesarean section, either emergent or elective.

Exclusion Criteria:

* History of myometrial intervention, such as myomectomy.
* History of genetic or acquired conditions that alter the anatomy of the uterus.
* History of coagulation disorders.
* History of connective tissue disorders, such as Lupus and Scleroderma, which may affect healing.
* Hemodynamically unstable patients due to a clinical condition prior to performing the cesarean section.
* Failure to sign the informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of uterine wall defect at the scar site | 6 to 16 weeks post-hysterotomy
  Performed via transvaginal ultrasound by a gynecologist trained in ultrasound who is blinded to the intervention

SECONDARY OUTCOMES:
Residual myometrial thickness of the uterine wall defect at the scar site | 6 to 16 weeks post-hysterotomy
  Performed via transvaginal ultrasound by a gynecologist trained in ultrasound who is blinded to the intervention
Myometrial thickness in the portion immediately cephalad to the residual myometrial defect | 6 to 16 weeks post-hysterotomy
  Performed via transvaginal ultrasound by a gynecologist trained in ultrasound who is blinded to the intervention
Myometrial thickness in the portion immediately caudal to the residual myometrial defect | 6 to 16 weeks post-hysterotomy
  Performed via transvaginal ultrasound by a gynecologist trained in ultrasound who is blinded to the intervention
Size of the uterine wall defect | 6 to 16 weeks post-hysterotomy
  Performed via transvaginal ultrasound by a gynecologist trained in ultrasound who is blinded to the intervention
Depth of the defect in the uterine wall | 6 to 16 weeks post-hysterotomy
  Performed via transvaginal ultrasound by a gynecologist trained in ultrasound who is blinded to the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Albaro J. Nieto, M.D., Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundación Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual patient data (IPD), since we are not allowed to share information concerning medical history of our patients or health workers.

REFERENCES:
- [Background] Betran AP, Ye J, Moller AB, Zhang J, Gulmezoglu AM, Torloni MR. The Increasing Trend in Caesarean Section Rates: Global, Regional and National Estimates: 1990-2014. PLoS One. 2016 Feb 5;11(2):e0148343. doi: 10.1371/journal.pone.0148343. eCollection 2016. PMID 26849801
- [Background] Buca D, Liberati M, Cali G, Forlani F, Caisutti C, Flacco ME, Manzoli L, Familiari A, Scambia G, D'Antonio F. Influence of prenatal diagnosis of abnormally invasive placenta on maternal outcome: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2018 Sep;52(3):304-309. doi: 10.1002/uog.19070. Epub 2018 Jul 29. PMID 29660186
- [Background] Silver RM, Fox KA, Barton JR, Abuhamad AZ, Simhan H, Huls CK, Belfort MA, Wright JD. Center of excellence for placenta accreta. Am J Obstet Gynecol. 2015 May;212(5):561-8. doi: 10.1016/j.ajog.2014.11.018. Epub 2014 Nov 20. PMID 25460838
- [Background] Palacios-Jaraquemada JM. Placental adhesive disorders, 1st ed. Berlin: DeGruyter editors, 2012 161 pages. ISBN 978-3-11-028238-2.
- [Background] Jauniaux E, Collins S, Burton GJ. Placenta accreta spectrum: pathophysiology and evidence-based anatomy for prenatal ultrasound imaging. Am J Obstet Gynecol. 2018 Jan;218(1):75-87. doi: 10.1016/j.ajog.2017.05.067. Epub 2017 Jun 24. PMID 28599899
- [Background] Vervoort AJ, Uittenbogaard LB, Hehenkamp WJ, Brolmann HA, Mol BW, Huirne JA. Why do niches develop in Caesarean uterine scars? Hypotheses on the aetiology of niche development. Hum Reprod. 2015 Dec;30(12):2695-702. doi: 10.1093/humrep/dev240. Epub 2015 Sep 25. PMID 26409016
- [Background] Fabres C, Aviles G, De La Jara C, Escalona J, Munoz JF, Mackenna A, Fernandez C, Zegers-Hochschild F, Fernandez E. The cesarean delivery scar pouch: clinical implications and diagnostic correlation between transvaginal sonography and hysteroscopy. J Ultrasound Med. 2003 Jul;22(7):695-700; quiz 701-2. doi: 10.7863/jum.2003.22.7.695. PMID 12862268
- [Background] Kremer TG, Ghiorzi IB, Dibi RP. Isthmocele: an overview of diagnosis and treatment. Rev Assoc Med Bras (1992). 2019 Jun 3;65(5):714-721. doi: 10.1590/1806-9282.65.5.714. PMID 31166450
- [Background] Sung S, Mikes BA, Martingano DJ, Mahdy H. Cesarean Delivery. 2024 Dec 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK546707/ PMID 31536313
- [Background] Dodd JM, Anderson ER, Gates S, Grivell RM. Surgical techniques for uterine incision and uterine closure at the time of caesarean section. Cochrane Database Syst Rev. 2014 Jul 22;2014(7):CD004732. doi: 10.1002/14651858.CD004732.pub3. PMID 25048608
- [Background] Cunningham FG, Larry C Gilstrap III, Hauth JC, Leveno KJ, Wenstrom KD, Gant NF. Obstetricia de Williams. Editorial Mac Graw Hill; 2019.
- [Background] Shao Y, Pradhan M. Higher Incision at Upper Part of Lower Segment Caesarean Section. JNMA J Nepal Med Assoc. 2014 Apr-Jun;52(194):764-70. PMID 26905701
- [Background] Armstrong F, Mulligan K, Dermott RM, Bartels HC, Carroll S, Robson M, Corcoran S, Parland PM, Brien DO, Brophy D, Brennan DJ. Cesarean scar niche: An evolving concern in clinical practice. Int J Gynaecol Obstet. 2023 May;161(2):356-366. doi: 10.1002/ijgo.14509. Epub 2022 Nov 21. PMID 36317541
- [Background] Monteagudo A, Carreno C, Timor-Tritsch IE. Saline infusion sonohysterography in nonpregnant women with previous cesarean delivery: the "niche" in the scar. J Ultrasound Med. 2001 Oct;20(10):1105-15. doi: 10.7863/jum.2001.20.10.1105. PMID 11587017
- [Background] Hofmeyr GJ, Mathai M, Shah A, Novikova N. Techniques for caesarean section. Cochrane Database Syst Rev. 2008 Jan 23;2008(1):CD004662. doi: 10.1002/14651858.CD004662.pub2. PMID 18254057
- [Background] Marotta ML, Donnez J, Squifflet J, Jadoul P, Darii N, Donnez O. Laparoscopic repair of post-cesarean section uterine scar defects diagnosed in nonpregnant women. J Minim Invasive Gynecol. 2013 May-Jun;20(3):386-91. doi: 10.1016/j.jmig.2012.12.006. Epub 2013 Jan 26. PMID 23357466
- [Background] Bij de Vaate AJ, van der Voet LF, Naji O, Witmer M, Veersema S, Brolmann HA, Bourne T, Huirne JA. Prevalence, potential risk factors for development and symptoms related to the presence of uterine niches following Cesarean section: systematic review. Ultrasound Obstet Gynecol. 2014 Apr;43(4):372-82. doi: 10.1002/uog.13199. PMID 23996650
- [Background] Palacios Jaraquemada JM, Garcia Monaco R, Barbosa NE, Ferle L, Iriarte H, Conesa HA. Lower uterine blood supply: extrauterine anastomotic system and its application in surgical devascularization techniques. Acta Obstet Gynecol Scand. 2007;86(2):228-34. doi: 10.1080/00016340601089875. PMID 17364288
- [Background] Dosedla E, Calda P. Can the final sonographic assessment of the cesarean section scar be predicted 6 weeks after the operation? Taiwan J Obstet Gynecol. 2016 Oct;55(5):718-720. doi: 10.1016/j.tjog.2015.07.006. PMID 27751422
- [Background] Gupta T, Singal K, Gupta N, Kohli S, Kanyal M. Comparative Study of USG and MRI in Evaluation of Isthmocele. J Obstet Gynaecol India. 2021 Jun;71(3):292-296. doi: 10.1007/s13224-021-01433-w. Epub 2021 Feb 17. PMID 34408349
- [Background] Savukyne E, Machtejeviene E, Paskauskas S, Ramoniene G, Nadisauskiene RJ. Transvaginal Sonographic Evaluation of Cesarean Section Scar Niche in Pregnancy: A Prospective Longitudinal Study. Medicina (Kaunas). 2021 Oct 12;57(10):1091. doi: 10.3390/medicina57101091. PMID 34684128
- [Background] Chen HY, Chen SJ, Hsieh FJ. Observation of cesarean section scar by transvaginal ultrasonography. Ultrasound Med Biol. 1990;16(5):443-7. doi: 10.1016/0301-5629(90)90166-a. PMID 2238250
- [Background] Tower AM, Frishman GN. Cesarean scar defects: an underrecognized cause of abnormal uterine bleeding and other gynecologic complications. J Minim Invasive Gynecol. 2013 Sep-Oct;20(5):562-72. doi: 10.1016/j.jmig.2013.03.008. Epub 2013 May 14. PMID 23680518
- [Background] Jauniaux E, Jurkovic D, Hussein AM, Burton GJ. New insights into the etiopathology of placenta accreta spectrum. Am J Obstet Gynecol. 2022 Sep;227(3):384-391. doi: 10.1016/j.ajog.2022.02.038. Epub 2022 Mar 3. PMID 35248577
- [Background] Khong TY. The pathology of placenta accreta, a worldwide epidemic. J Clin Pathol. 2008 Dec;61(12):1243-6. doi: 10.1136/jcp.2008.055202. Epub 2008 Jul 19. PMID 18641410
- [Background] Tantbirojn P, Crum CP, Parast MM. Pathophysiology of placenta creta: the role of decidua and extravillous trophoblast. Placenta. 2008 Jul;29(7):639-45. doi: 10.1016/j.placenta.2008.04.008. Epub 2008 Jun 2. PMID 18514815
- [Background] Abdallah W, Najib B, Atallah D. The higher incision at upper part of lower uterine segment in caesarean section can decrease the incidence of placenta accreta spectrum. Med Hypotheses. 2020 Nov;144:110228. doi: 10.1016/j.mehy.2020.110228. Epub 2020 Sep 2. PMID 33254537
- [Background] Vikhareva O, Rickle GS, Lavesson T, Nedopekina E, Brandell K, Salvesen KA. Hysterotomy level at Cesarean section and occurrence of large scar defects: a randomized single-blind trial. Ultrasound Obstet Gynecol. 2019 Apr;53(4):438-442. doi: 10.1002/uog.20184. PMID 30484920
- [Background] Hayakawa H, Itakura A, Mitsui T, Okada M, Suzuki M, Tamakoshi K, Kikkawa F. Methods for myometrium closure and other factors impacting effects on cesarean section scars of the uterine segment detected by the ultrasonography. Acta Obstet Gynecol Scand. 2006;85(4):429-34. doi: 10.1080/00016340500430436. PMID 16612704
- [Background] Hamar BD, Saber SB, Cackovic M, Magloire LK, Pettker CM, Abdel-Razeq SS, Rosenberg VA, Buhimschi IA, Buhimschi CS. Ultrasound evaluation of the uterine scar after cesarean delivery: a randomized controlled trial of one- and two-layer closure. Obstet Gynecol. 2007 Oct;110(4):808-13. doi: 10.1097/01.AOG.0000284628.29796.80. PMID 17906013
- [Background] Yazicioglu F, Gokdogan A, Kelekci S, Aygun M, Savan K. Incomplete healing of the uterine incision after caesarean section: Is it preventable? Eur J Obstet Gynecol Reprod Biol. 2006 Jan 1;124(1):32-6. doi: 10.1016/j.ejogrb.2005.03.023. Epub 2005 Jul 14. PMID 16023780
- [Background] Yilmaz Baran S, Kalayci H, Dogan Durdag G, Yetkinel S, Alemdaroglu S, Cok T, Bulgan Kilicdag E. Single- or double-layer uterine closure techniques following cesarean: A randomized trial. Acta Obstet Gynecol Scand. 2021 Mar;100(3):531-537. doi: 10.1111/aogs.14018. Epub 2020 Oct 30. PMID 33029804
- [Background] Roberge S, Demers S, Girard M, Vikhareva O, Markey S, Chaillet N, Moore L, Paris G, Bujold E. Impact of uterine closure on residual myometrial thickness after cesarean: a randomized controlled trial. Am J Obstet Gynecol. 2016 Apr;214(4):507.e1-507.e6. doi: 10.1016/j.ajog.2015.10.916. Epub 2015 Nov 11. PMID 26522861
- [Background] Jaki T, Vasileiou D. Factorial versus multi-arm multi-stage designs for clinical trials with multiple treatments. Stat Med. 2017 Feb 20;36(4):563-580. doi: 10.1002/sim.7159. Epub 2016 Nov 2. PMID 27804166
- [Background] Saccone G, De Angelis MC, Zizolfi B, Gragnano E, Musone M, Zullo F, Bifulco G, Di Spiezio Sardo A. Monofilament vs multifilament suture for uterine closure at the time of cesarean delivery: a randomized clinical trial. Am J Obstet Gynecol MFM. 2022 May;4(3):100592. doi: 10.1016/j.ajogmf.2022.100592. Epub 2022 Feb 4. PMID 35131497